CLINICAL TRIAL: NCT00473460
Title: A Double-blind, Randomized, Placebo-controlled Study to Investigate Chronic Intermittent-pulse-therapy of Moxifloxacin as a Prevention of Acute in Exacerbation Out-patients With Chronic Bronchitis.
Brief Title: Intermittent Moxifloxacin Therapy For The Prevention Of Acute Exacerbations In Patients With Chronic Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11229; EudraCT No: 2004-000404-40
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Lung Diseases; Bronchitis, Chronic
Keywords: Chronic bronchitis; Chronic obstructive pulmonary disease; Acute exacerbation of chronic bronchitis; Prevention therapy; Antibiotics; Fluoroquinolone; Moxifloxacin; AECB
MeSH Terms: conditions — Lung Diseases; Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Avelox (Moxifloxacin, BAY12-8039), 400 mg capsules orally once daily for 5 days every 8 weeks
  Arms: Arm 1
Drug: Placebo — Matching placebo capsules orally once daily for 5 days every 8 weeks.
  Arms: Arm 2

SUMMARY:
Moxifloxacin, is being tested at approximately 60 study centres in 15 countries to determine if this drug, when taken periodically in addition to the patients normal treatment, is effective at reducing the number of flare-ups of chronic bronchitis he has. Approximately 1132 subjects will participate, and it is expected that the study will run for 2 years in order to reach that goal. The patients individual involvement in the study will be 17 months. Moxifloxacin will be compared to a placebo drug (no active ingredients). The study medication (moxifloxacin or placebo) will be taken in addition to the patients normal medication for chronic bronchitis. In addition to the first clinic visit, called a screening visit, the patient will be required to come back to the clinic for ten more study visits, every 8 weeks. At the first visit the study co-ordinator will provide him with the dates for all the visits. Over a period of 48 weeks the patient will return to the clinic on 6 occasions where he will receive the study medication which he will take for five days, in addition to his normal treatment for chronic bronchitis. After this time the patient will enter a follow up period for 24 weeks, where he will come to the clinic for assessments and continue to take his normal medication but not receive the study drug. A complete medical history will be taken at the first visit, including the patients past and current smoking habit. A breath test will be performed to assess how well his lungs are functioning. In addition, he will also be asked to provide a sputum sample for a microbiological examination to identify any bacteria present in the sample. The patient must be able to provide a sputum sample at the screening visit. If the patient meets all the inclusion / exclusion criteria for the study, he will be allocated randomly to one of the following treatment groups at the second visit.- Treatment group 1: Receives moxifloxacin orally once daily for five days.- Treatment group 2: Receives a matching placebo once daily for five days.In between each visit (four weeks after your clinic visit), the study site co-ordinator will contact the patient to check on his well being. If the patient or the doctor decides to stop the patients participation in the trial for any reason, the patient will be required to return to the clinic for a physical examination, take a breath test, provide a sputum sample (if possible) and have a blood sample taken.

ELIGIBILITY:
Inclusion Criteria:

* Male or female out-patients >/= 45 years
* Subjects suffering from chronic bronchitis
* FEV1</= 70% and FEV1/FVC </= 70% predicted from age, height and sex
* No documented episode of AECB (requiring treatment) within 6 weeks of randomization and not experiencing an exacerbation at the time of screening
* Sputum production on most days, even when exacerbation free
* Subjects presented with at least two documented (i.e. requiring antibiotics and/or systemic steroid administration) acute exacerbation episodes during the last 12 monthsIf receiving chronic therapy with inhaled long acting bronchodilators and/or inhaled or systemic steroids, the treatment must have remained stable for the preceding 6 weeks prior to screening
* Smoking history of at least 20 pack-years
* Subjects willing and able to give fully informed written consent

Exclusion Criteria:

* Subjects with contra-indications to moxifloxacin- Known bronchial carcinoma, pulmonary tuberculosis, cystic fibrosis, documented chronic bronchial asthma or diffuse bronchiectasis- Subjects who are actively participating in intensive pulmonary rehabilitation programs
* Subjects with a known history of chronic colonization of pathogenic organisms resistant to moxifloxacin, e.g. Pseudomonas spp, MRSA
* No systemic or inhaled antibiotic therapy during the 6 weeks prior to screening and any long term antibiotic usage
* Subjects requiring home ventilatory support for COPD and those who have a tracheostomy in situ (subjects requiring home/potable oxygen therapy or CPAP for sleep apnea can be included)

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1404 (Actual)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations after 48 weeks of intermittent pulse treatment | After 48 weeks of treatment

SECONDARY OUTCOMES:
Impact of treatment on the health related Quality of Life in St. George's Respiratory Questionaire (SGRQ) scores | At week 48
Deterioration in lung function test (PFEV1) | At week 48
Frequency of hospitalisation | At week 48
Mortality rates | At week 48
Time of first exacerbation | Through to week 48
Frequency of acute exacerbation of chronic bronchitis | At week 24 and 72 (end of follow-up)
Time to next exacerbation from last pulsed dose | At week 48
Length of exacerbations | Through to week 48
Percentage of exacerbation free time | Through to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (63):
- United States (10):
  - Tucson, Arizona
  - Long Beach, California
  - Los Angeles, California
  - Bay Pines, Florida
  - Kansas City, Missouri
  - Buffalo, New York
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
- Les Escaldes, Andorra
- Argentina (2):
  - San Juan Bautista, Buenos Aires
  - Buenos Aires, Buenos Aires F.D.
- Brazil (3):
  - Juiz de Fora, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Chile (2):
  - Santiago
  - Valparaíso
- France (6):
  - Arras
  - Mont-de-Marsan
  - Nice
  - Orthez
  - Rosiers-d'Égletons
  - Strasbourg
- Germany (9):
  - Kaufbeuren, Bavaria
  - Hamburg, Hamburg
  - Gelnhausen, Hesse
  - Hanover, Lower Saxony
  - Rotenburg (Wümme), Lower Saxony
  - Witten, North Rhine-Westphalia
  - Neuwied, Rhineland-Palatinate
  - Bad Segeberg, Schleswig-Holstein
  - Berlin, State of Berlin
- Greece (2):
  - Rio, Patras
  - Athens
- Ireland (2):
  - Dublin, Dublin
  - Dublin
- Israel (4):
  - Afula, Israel
  - Ashkelon, Israel
  - Bat Yam, Israel
  - Tel Aviv, Israel
- Italy (3):
  - Ferrara
  - Milan
  - Pavia
- Mexico (3):
  - Chihuahua City, Chihuahua
  - Guadalajara, Jalisco
  - Mérida, Yucatán
- South Africa (6):
  - Bloemfontein, Free State
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
  - Paarl, Western Cape
- Spain (6):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Ronda, Málaga
  - Valencia, Valencia
  - Valladolid, Valladolid
- United Kingdom (4):
  - Bristol, Avon
  - London, Greater London
  - Birmingham, West Midlands
  - Leeds, West Yorkshire

REFERENCES:
- [Derived] Sethi S, Jones PW, Theron MS, Miravitlles M, Rubinstein E, Wedzicha JA, Wilson R; PULSE Study group. Pulsed moxifloxacin for the prevention of exacerbations of chronic obstructive pulmonary disease: a randomized controlled trial. Respir Res. 2010 Jan 28;11(1):10. doi: 10.1186/1465-9921-11-10. PMID 20109213
- See also: Click here and search for information on EMA — http://www.clinicaltrialsregister.eu